CLINICAL TRIAL: NCT00233090
Title: Post-TBI Fatigue and Its Treatment
Brief Title: Post-Traumatic Brain Injury (Post-TBI) Fatigue and Its Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO #02-0677; H133A020501
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Fatigue
Keywords: Fatigue; TBI; brain injury; Modafinil; traumatic brain injury
MeSH Terms: conditions — Fatigue; Brain Injuries; Brain Injuries, Traumatic | interventions — Modafinil

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Modafinil (Experimental): single dose of 200 mg. a day of modafinil for four weeks
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — single dose of 200 mg. a day of modafinil for four weeks
  Arms: Modafinil
Drug: Placebo — daily dose of placebo for four weeks.
  Arms: Placebo

SUMMARY:
Randomized clinical trial of modafinil vs. placebo for treatment of fatigue after TBI.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to examine the efficacy of the drug modafinil as a treatment for fatigue post TBI.

Background: After TBI, fatigue is one of the most common complaints, as documented in our work and that of many other researchers. People with TBI experience fatigue that seems to them out of proportion to whatever work they are doing or effort they are making. Fatigue after TBI is associated with decreased participation in normal activities in the community and has been linked to depression.

Need for Research: Research on use of drugs to treat post-TBI fatigue is inadequate. While studies of fatigue in people with other chronic conditions suggest that modafinil helps relieve fatigue and has fewer side effects than some other drugs used in treating fatigue, the use of modafinil has not yet been tested in people with TBI.

Current and Future Research Activity: More than 100 men and women volunteers who complain of post-TBI fatigue will be randomly assigned to a 4-week period of taking modafinil or a placebo. At the beginning and end of the study, the severity of their fatigue and associated symptoms (e.g., cognitive function, mood, pain, daytime sleepiness, sleep quality, health status) will be assessed, as well as their participation in activities and perceived quality of life. It is hypothesized that modafinil will reduce the symptoms of fatigue and will increase level of activity and perceived quality of life to a significantly greater extent than will the placebo.

ELIGIBILITY:
Inclusion Criteria:

- Individuals who sustained a TBI with a documented loss of consciousness or evidence of a TBI on neuroimaging studies and who are at least 12 months post-injury, who complain of fatigue and who have scores of 22 or above on the Barroso Fatigue Scale will be eligible to participate in this study. Subjects must not meet criteria for alcohol or substance abuse using the Structured Clinical Interview for DSM-IV (SCID) for at least six months prior to study enrollment.

Exclusion Criteria:

- Diagnosis of chronic neurological disease (including Lyme disease), narcolepsy, current infectious disease, chronic fatigue syndrome, fibromyalgia, anemia, hypothyroidism not adequately controlled with medication, blood pressure greater 150/100 mm Hg, or clinically significant major systemic disease. In addition, individuals taking medications which are known to cause fatigue will be excluded from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne A Gordon, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12) | 54 (13) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: Self-report of fatigue
Time Frame: comparison pre and post treatment
Population: Study terminated due to low enrollment. data was not analyzed and is no longer available for analysis. Data not kept electronically and study records are no longer available.
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cognitive Performance
Description: Cognitive performance
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mood
Description: mood
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain
Description: pain
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Sleep Quality
Description: sleep quality
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Health Status
Description: health status
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Participation
Description: participation
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Quality of Life
Description: quality of life
Time Frame: comparison pre and post treatment
Population: as for outcome 1
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

LIMITATIONS AND CAVEATS:
Study was terminated due to insufficient recruitment. Data analysis not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes